CLINICAL TRIAL: NCT01060085
Title: A Comparison of the Diagnostic Accuracy of Adjunctive Digital Breast Tomosynthesis Versus Adjunctive Contrast Enhanced Breast Magnetic Resonance Imaging in the Preoperative Assessment of Breast Cancer
Brief Title: Digital Breast Tomosynthesis Versus Contrast Enhanced Magnetic Resonance Imaging (MRI) for Breast Cancer Staging
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D0842
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ductal Carcinoma In Situ; Invasive Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast Cancer: Women shown to have DCIS or invasive breast cancer by fine needle aspiration cytology and/or core needle biopsy.

SUMMARY:
The primary objective of this study is to compare the diagnostic accuracy of Digital Breast Tomosynthesis (DBT) versus that of Contrast Enhanced Magnetic Resonance Imaging (CEMRI) in determining the size of breast cancer preoperatively.

Secondary objectives include:

1. Comparing the operating characteristics of each combined imaging protocol with respect to the reference standard, i.e. histopathologic assessment, of additional non-index lesions.
2. Comparison of re-excision rates based on estimated disease extent from adjunctive CEMRI vs. adjunctive DBT.
3. Evaluation of patient satisfaction with regard to the adjunctive modality (DBT vs. CEMRI).

DETAILED DESCRIPTION:
STUDY OVERVIEW

Subjects are enrolled within 4 weeks of the date of diagnosis of biopsy proven ductal carcinoma in-situ (DCIS) or Invasive Breast Cancer. Approximately 50 subjects will be enrolled. In addition to Dartmouth-Hitchcock Medical Center's (DHMC)current standard imaging practice, i.e. bilateral mammography with or without sonography and bilateral CEMRI, all subjects will undergo bilateral DBT within four weeks of CEMRI and prior to surgical treatment. Usual clinical practice, i.e. interpretation of current standard imaging (Mammography, Sonography and CEMRI), and clinical assessment based on physical exam as well, as discussion with the patient and breast surgeon of record, will dictate local treatment, i.e. surgical excision only, breast conservation therapy (BCT) or mastectomy.

Any routine diagnostic examinations completed as part of the subject's standard of care imaging will be read and interpreted as part of the patient's standard of care. There will be no delays in reading or interpretation of the routine care images.

Blinded reads of the DBT and CEMRI images will be conducted, with the patient's mammography +/- sonography available for reference. The interpreting radiologists ("readers") will evaluate tumor size and extent of disease, along with the presence or absence of multi-focality or contralateral disease. The two imaging paradigms will be compared in the estimation of breast cancer extent using the gold-standard histologic result.

DBT mammography may provide new or different information about the index lesion than standard imaging, but this will not alter clinical management. However, if DBT detects an additional abnormality separate from the index lesion either in the ipsilateral or contralateral breast, it will be evaluated further with standard imaging technology (e.g. diagnostic mammography and or sonography) targeted to this site to assess the level of suspicion for malignancy and potential need for biopsy.

PROCEDURES

Tomosynthesis Acquisition

Study participants shown to have DCIS or invasive breast cancer by fine needle aspiration cytology and/or core needle biopsy, and who have signed informed consent, will undergo a bilateral DBT mammogram within 4 weeks of CEMRI (prior to surgical treatment). The DBT mammogram includes a 2D acquisition and a 3D acquisition, under the same compression in both the standard craniocaudal (CC) and mediolateral (MLO) projections. In the rare instance that the index malignancy is not included on a view due to a chest wall location, a single repeat view of the involved (i.e. cancerous) breast will be performed in an attempt to image the malignancy on the combined DBT mammogram. For each view, the subject will be positioned and compressed as for standard mammographic imaging. The patient will remain under compression for no more than 15 seconds. During the compression, a 3D dataset (about a 4 second exposure) and a 2D dataset (about a 2 second exposure) will be acquired. Once the subject is positioned and compressed, the technologist will activate the motion of the x-ray tube to move to the starting position of -7.5 degrees. The technologist will then start the tomosynthesis 3D acquisition, which is completed at +7.5 degrees (an arc of 15 degrees). The x-ray tube then by design moves back to the center and automatically acquires the 2D dataset. At the conclusion of image acquisition, the compression is automatically released.

A Radiologic Technologist registered for radiography and mammography will perform the tomosynthesis study. The technologist performing the DBT exam has been trained in the use and operation of the DBT imaging system.

Device Description

A DBT system similar to the commercially available product ('Selenia Dimensions', Hologic, Inc., Danbury CT) will be used for the data collection. The 'Selenia Dimensions' 2D/3D digital mammography system has been approved by the FDA for screening and diagnostic breast imaging.

The breast tomosynthesis system is a digital mammography system (Hologic, Inc, Danbury, CT) that is capable of producing standard two-dimensional images and a three-dimensional tomosynthesis mammogram. The 2D and 3D tomographic datasets are acquired under the same compression. The breast tomosynthesis system employs a tungsten target anode with interchangeable rhodium, silver, and aluminum x-ray filters. The filtration material is chosen based on breast thickness and exam protocol and, along with the tungsten target, minimizes x-ray dose while maximizing image content. The three-dimensional tomosynthesis x-ray imaging technology involves acquiring images of a stationary compressed breast, at multiple angles during a short-scan. The individual images are then reconstructed into a series of thin high-resolution slices that are displayed individually or in a dynamic cine mode. When in combination mode, the system acquires both the 3D dataset and then the 2D standard mammographic image. The dose for a single combination 2D/3D acquisition for the "average breast" i.e. compressed breast thickness of 4.5 cm, 50% fat, 50% glandular composition is approximately 2.45 mGy, less than the FDA limit for a single mammogram image (3 mGy) for the same breast thickness and composition.

The DBT system will only be used for subjects who have signed the Informed Consent.

Quality Control

The Hologic Tomosynthesis Digital Mammography System (DBT) will be checked by a qualified medical physicist prior to any testing or imaging of subjects to assure the system is operating correctly with optimum image quality. A Study Technologist will review images, obtain phantom images and check system operation on a periodic basis to assure that optimum image quality is maintained. The quality control procedures described in the systems' operator manuals will be used throughout the trial. If there is any noticeable degradation in image quality, a Hologic engineer will be called immediately to recalibrate or repair the system.

CEMRI

Each subject will undergo bilateral CEMRI as part of usual clinical practice, not because of their participation in the study. Subjects who are unable to undergo contrast enhanced MRI due to contraindications to MRI or gadolinium based intravenous contrast are not eligible for study enrollment.

Image Interpretation

The DBT images will be evaluated by a Mammography Quality Standards Act certified radiologist. There will be two readers for each subject: one reader will interpret DBT (blinded to results of CEMRI), while the second reader will interpret CEMRI (blinded to results of DBT). Each reader interprets the adjunct exam (i.e. DBT or CEMRI) unblinded to conventional imaging (i.e. mammography +/- sonography) and completes the appropriate rating instrument.

Size Determination

Study Readers will estimate the maximal in plane diameter in at least two imaging planes of the index malignant lesion. For DBT, maximal diameters should be measured in the CC and MLO projections. For CEMRI, maximal diameters should be measured in axial and sagittal projections. Readers will also report on and diagram the location of additional lesions that are not considered definitely benign.

Histological Interpretation

The specimen (lumpectomy or mastectomy) is sequentially sectioned into 5 mm slices and the number of slices is recorded in the gross description. Targeted sections are taken of both lumpectomies and mastectomies by sampling lesions identified by imaging (per usual clinical protocol). Such lesions are submitted as appropriate along with 1-2 sections of a surrounding cuff of normal appearing parenchyma in each appropriate direction. The distance between multiple lesions is measured, and in such cases a single section of intervening tissue is submitted for histologic examination. Incidental lesions identified on gross exam are sampled as appropriate. The histopathologic specimen is viewed by a pathologist with 3-20 years of experience in breast pathology. Invasive disease is graded according to the Nottingham Bloom Scarff Richardson system. DCIS is graded according to a modified Van Nuys system, including the nuclear grade, the presence or absence of necrosis, and the pattern of growth. The number of consecutive slides containing DCIS will be multiplied by the approximate thickness of each tissue section (5mm) in order to determine the histopathologic size.

Tumor size will be determined by gross examination of the pathology specimen when visible on gross examination. Tumor size estimate in this case will reflect an aggregate of invasive and non-invasive, i.e. DCIS, components.

If no gross lesion is seen, the measurement of tumor size will be determined by the microscopic measurement of the lesion. Since the 2 components are intermingled, the size reported represents an aggregate size.

In addition to the gross exam measurement, if a lesion is substantially composed of DCIS, (i.e. extensive intraductal component present) by microscopic examination, we will specify the size of both the invasive component (by microscopic exam) as well as a measurement of the DCIS component (by microscopic exam) and provide an aggregate size of both invasive and DCIS components).

In cases of invasive cancer with an extensive component of DCIS treated with mastectomy or a very wide local excision, standard pathologic sampling of the lesion may not allow for accurate microscopic size estimate of the lesion. In these select cases the pathologist will indicate the type of growth pattern of the DCIS component as either "mass-like" or "non mass-like".

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity
* Subject is at least 30 years old
* Subject has histologically proven DCIS or invasive breast carcinoma.
* Subject is able to undergo CEMRI at DHMC-Lebanon

Exclusion Criteria:

* Patients who are pregnant or think they may be pregnant
* Patients who are breast-feeding.
* Patients who have significant existing breast trauma
* Subjects unable or unwilling to undergo informed consent
* Absolute contraindication to CEMRI, including:

  1. presence of implanted electrical device (pacemaker or neurostimulator),aneurysm clip, or metallic foreign body in or near the eyes
  2. life threatening allergy to gadolinium contrast
* CEMRI performed at institution other than DHMC Lebanon
* Patients undergoing neoadjuvant therapy
* Patients with maximum tumor diameter >5cm
* Patients presenting with Inflammatory Breast Cancer
* Patients with gross axillary lymphadenopathy on clinical exam or by imaging
* Maximum breast size limitation: i.e. breast size that exceeds the size of the large format image receptor (24cm x 29cm) on any view

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have histologically proven, non-inflammatory, breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2009-02; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison between the accuracy of DBT vs. CEMRI using two measurements: 1. Maximal diameter estimate by imaging modality and 2. Maximal diameter based on histopathology gold standard. | surgical pathology results completed

SECONDARY OUTCOMES:
True positives, true negatives, false positives and false negatives for: 1. Multi-focality defined as additional discrete discontinuous tumor foci that are at least 2.5 cm separate from the index lesion. 2. Contralateral disease: presence/absence | surgical pathology results completed
Predicted re-excision rates based on size estimates from each imaging paradigm | surgical pathology results completed
Patient satisfaction survey for DBT and CEMRI imaging | patient completion of DBT and CEMRI imaging

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Poplack, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No